CLINICAL TRIAL: NCT07002320
Title: ASpiRE: A Proof-of-mechanism and Proof-of-concept Clinical Trial Evaluating the Safety, Tolerability, Biological and Anti-tumour Activity of Apalutamide With Dual CXCR1 and CXCR2 Blockade by SX-682 for Men Suffering From Metastatic Castration-resistant Prostate Cancer (mCRPC)
Brief Title: Investigating SX-682 in Combination With Apalutamide in Metastatic Castration-resistant Prostate Cancer
Acronym: ASpiRE
Status: Recruiting | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Institute of Cancer Research, United Kingdom (Other)
Collaborators: Prostate Cancer UK (Other); Janssen Pharmaceutica N.V., Belgium (Industry); Oncology Institute of Southern Switzerland (Other); Syntrix Biosystems, Inc. (Industry); Royal Marsden NHS Foundation Trust (Other); Cambridge University Hospitals NHS Foundation Trust (Other); Belfast Health and Social Care Trust (Other); Institute of Oncology Research (IOR) (Unknown)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: CCR6041; 1008729 (Registry Identifier: Integrated Research Application System (IRAS))
Record Dates: First submitted 2025-05-06; First posted 2025-06-03 (Actual); Last update posted 2025-12-04 (Actual); Status verified 2025-12

CONDITIONS: Metastatic Castrate-Resistant Prostate Cancer (mCRPC)
Keywords: Prostate cancer
MeSH Terms: conditions — Prostatic Neoplasms | interventions — apalutamide

STUDY DESIGN:
Intervention Model Description: Phase 1 will use a 3+3 design to investigate escalating doses of SX-682 in combination with Apalutamide.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Phase I: Dose Escalation (Experimental): Phase I will identify a biologically active and tolerable (safe) dose range of SX-682 in combination with Apalutamide in patients with metastatic castrate-resistant prostate cancer (mCRPC).
  Interventions: Drug: SX-682; Drug: Apalutamide
- Phase II: Dose Expansion (Experimental): Phase I will investigate the anti-tumour activity of tolerable doses of SX-682 in combination with Apalutamide in patients with metastatic castrate-resistant prostate cancer (mCRPC). Patients will be treated at dose levels deemed to be tolerable and biologically active, based on safety and efficacy data from Dose Escalation.
  Interventions: Drug: SX-682; Drug: Apalutamide

INTERVENTIONS:
Drug: SX-682 — SX-682 is supplied as 100mg film coated tablets.
Drug: Apalutamide — Apalutamide is supplied as 60mg film coated tablets.

SUMMARY:
ASpiRE will investigate the effect of the drug SX-682 in combination with Apalutamide in men suffering from metastatic castration-resistant prostate cancer (mCRPC).

ELIGIBILITY:
Inclusion Criteria:

1. Written informed consent and be capable of cooperating with treatment.
2. Age ≥ 18 years.
3. Histologically or biochemically confirmed adenocarcinoma of the prostate and with tumour tissue accessible for research analysis for this trial. Patients who have no histological diagnosis must be willing to undergo a biopsy to prove prostate adenocarcinoma.
4. Patients recruited to phase 1 dose escalation cohorts must have biopsiable disease and consent to mandatory pre- and post-treatment biopsies (baseline and on Cycle 2 Day 1).
5. Metastatic castration-resistant prostate cancer.
6. All patients must have documented resistance to 1 prior next generation antiandrogen therapy (NAAT) defined as:

   For phase 1 and phase 2 Cohorts:

   Patients who have progressed after either enzalutamide, Apalutamide or darolutamide (having received a minimum of 12-weeks of enzalutamide, Apalutamide or darolutamide) will enter phase 1 or phase 2 cohorts directly. Patients that have previously received abiraterone but not an AR antagonist should receive a lead-in with Apalutamide on trial and receive the combination on progression through the lead-in.
7. Documented prostate cancer progression as assessed by the investigator with RECIST v1.1 and PCWG3 criteria (Section 3.5) with at least two of the following criteria:

   1. Progression of soft tissue/visceral disease by RECIST v1.1 and/or,
   2. Progression of bone disease by PCWG3 bone scan criteria and/or,
   3. Progression of PSA by PCWG3 PSA criteria.
8. PSA ≥ 10ng/ml.
9. Received prior castration by orchiectomy and/or ongoing luteinizing hormone releasing hormone agonist treatment.
10. Ongoing androgen deprivation with serum testosterone < 50 ng/dL (< 1.7 nM).
11. Eastern Cooperative Oncology Group (ECOG) Performance Status of ≤2.
12. Documented willingness to use an effective means of contraception while participating in the study and for 6 months post last treatment dose.
13. Able to swallow the study drug.
14. All efforts should be made to discontinue steroid usage but up-to 5mg BD prednisolone (or equivalent) will be allowed.
15. Haematological and biochemical indices within the ranges shown below. These measurements must be performed within one week (Day -7 to Day 1) before the patient goes on trial.

Haemoglobin (Hb) ≥ 9.0 g/dL Absolute neutrophil count ≥ 1.5 x 109/L Platelet count ≥ 100 x 109/L WBC ≥ 3.0 x 109/L Calculated creatinine clearance ≥ 50 mL/min (uncorrected value) Serum bilirubin ≤ 1.5 x upper limit of normal (ULN) unless documented Gilbert's disease., in which case ≤ 3 x ULN is permissible Alanine aminotransferase (ALT) and aspartate aminotransferase (AST) ≤ 2.5 x (ULN) unless raised due to known metastatic liver disease in which case ≤ 5 x ULN is permissible

Exclusion Criteria:

1. Surgery, chemotherapy, or other anti-cancer therapy within 4 weeks prior to trial entry/randomisation into the study (with the exception of abiraterone, enzalutamide, Apalutamide or darolutamide). Any other therapy for prostate cancer, other than gonadotropin releasing hormone analogue therapy, such as progesterone, medroxyprogesterone, progestins or 5-alpha reductase inhibitors, must be discontinued at least 2 weeks before the first dose of the study drug.
2. Participation in another interventional clinical trial of an IMP within 4 weeks prior to trial entry. Participation in trials of licensed medications is allowed provided the medication is not a prohibited concomitant medication.
3. Prior limited field radiotherapy within 2 weeks and wide field radiotherapy within 4 weeks prior to trial entry.
4. Clinical and/or biochemical evidence of hyperaldosteronism or hypopituitarism.
5. History of seizures or other predisposing factors including, but not limited to, underlying brain injury, stroke, primary brain tumours, brain metastases and leptomeningeal disease, or alcoholism.
6. Malabsorption syndrome or other condition that would interfere with enteral absorption.
7. Any of the following cardiac criteria:

   * QTcF interval > 470 msec.
   * Clinically important abnormalities including rhythm, conduction, or electrocardiogram (ECG) changes (left bundle branch block, third degree heart block).
   * Factors predisposing to QT prolongation including heart failure, hypokalaemia, congenital long QT syndrome, family history of prolonged QT syndrome, unexplained sudden death (under 40) and concomitant medications known to prolong QT interval.
   * Coronary artery bypass, angioplasty, vascular stent, myocardial infarction, angina, congestive heart failure (NYHA ≥ grade 2) i or transient ischaemic attack) in the last 6 months (see appendix 4 for NYHA scale).
   * Uncontrolled hypotension (systolic blood pressure < 90mmHg).
   * Uncontrolled hypertension on optimal medical management.
8. Clinically significant history of liver disease (Child-Pugh B or C, viral or other hepatitis, current alcohol abuse or cirrhosis).
9. Any other finding giving reasonable suspicion of a disease or condition that contraindicates the use of an investigational drug or that may affect interpretation of the results or renders the patients at high risk from treatment complications, e.g., patients with a hypersensitivity to the active substance or any of the excipients.
10. Malignancy other than prostate cancer within 5 years of trial entry except for adequately treated basal cell carcinoma.
11. Unresolved significant toxicity from prior therapy (except alopecia and grade 1 peripheral neuropathy).
12. Inability to comply with study and follow-up procedures.
13. Predominantly small cell or neuroendocrine differentiated (> 20% of cells) prostate cancer.
14. Immunocompromised patients.
15. Active or uncontrolled autoimmune disease requiring corticosteroid therapy.
16. History of thromboembolic disease within 12 months of commencement of trial.
17. At high-risk because of non-malignant systemic disease including active infection and any serious concurrent illness.
18. Any known intolerance to Apalutamide, SX-682, or to any constituents.
19. Symptoms of COVID-19 and/or documented COVID-19 infection.
20. Is taking any of the following prohibited medications:

    * Aminophylline/theophylline
    * Atypical antipsychotics (eg, clozapine, olanzapine, risperidone, ziprasidone)
    * Buproprion
    * Lithium
    * Meperidine and pethidine
    * Phenothiazine antipsychotics (eg, chlorpromazine, mesoridazine, thioridazine)
    * Tricyclic and tetracyclic antidepressants (eg, amitriptyline, desipramine, doxepin, imipramine, maprotiline, mirtazapine
    * Warfarin or coumarin-like anticoagulants
21. History of previous non-infectious pneumonitis requiring steroid treatment, or active non-infectious pneumonitis.
22. History of previous severe drug induced severe cutaneous reaction including but not limited to Steven-Johnson's syndrome/toxic epidermal necrolysis, drug reaction with eosinophilia and systemic symptoms (DRESS).

Min Age: 18 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Gender Based: Yes — Male
Enrollment: 78 (Estimated)
Dates: Start 2025-04-28 (Actual); Primary Completion 2029-10 (Estimated); Study Completion 2029-10 (Estimated)

PRIMARY OUTCOMES:
Biologically active and tolerable dose range | From start of treatment to end of Cycle 2 Day 1 (each cycle is 28 days)
  The biological active and tolerable combination doses are those that satisfy observed DLT rate<33% and demonstrate reduction in myeloid derived suppressor cells (MDSCs).
Anti-tumour activity of SX-682 when administered with Apalutamide | 24 months
  Response rate on the basis of Prostate Cancer Working Group 3 (PCWG3), and/or Response Evaluation Criteria in Solid Tumors (RECIST) v1.1 criteria.

SECONDARY OUTCOMES:
Safety and tolerability profile as assessed by Common Terminology Criteria for Adverse Events (CTCAE) v5.0 | 12 months
Steady state pharmacokinetic parameters (CSSmin and CSSMax) | At the end of Cycle 2 Day 1 (each cycle is 28 days).
Number of patients with Prostate Specific Antigen (PSA) decline greater than 50% | 24 months
Soft tissue objective response (CR or PR) by RECIST v1.1 | From date of enrolment until the date of first documented progression or date of death from any cause, whichever came first, assessed up to 36 months.
Changes in circulating tumour DNA (ctDNA) tumour fractions (TF). | 24 months
Progression free survival | From date of enrolment until the date of first documented progression or date of death from any cause, whichever came first, assessed up to 60 months
Overall survival | From date of enrolment to date of death from any cause, assessed up to 60 months.
Relative changes in circulating neutrophils | 24 months
Impact on quality of life using Brief Pain Inventory (BPI) Questionnaire | 24 months
  The BPI questionnaire assesses pain severity and impact of pain on daily functioning. Higher scores indicate greater pain severity and interference with daily life.
Impact of treatment toxicity using Functional Assessment of Chronic Illness Therapy (FACIT)-GP5 Questionnaire | 24 months
  Score between 0-4 with high score meaning patients are bothered by treatment side effects
Relative changes in intra-tumour myeloid derived suppressor cells (MDSCs) | 24 months

CONTACTS AND LOCATIONS:
Overall Officials: Professor Johann de Bono, MB ChB, FRCP, MSc, PhD, FMedSc, Study Director — Institute of Cancer Research, United Kingdom
Locations (4):
- Oncology Institute of Southern Switzerland, Bellinzona, Switzerland
- United Kingdom (3):
  - Belfast Health and Social Care Trust, Belfast
  - Cambridge University Hospitals NHS Foundation Trust, Cambridge
  - The Royal Marsden NHS Foundation Trust - Drug Development Unit, Sutton

IPD SHARING:
Plan to Share IPD: Undecided